CLINICAL TRIAL: NCT05369104
Title: A Pilot, Multicenter, Randomized, Non-Comparative, Double-Blind Study of Phage Therapy in Patients With Hip or Knee Prosthetic Joint Infection Due to Staphylococcus Aureus Treated With DAIR and Antibiotic Therapy.
Brief Title: Phage Therapy in Prosthetic Joint Infection Due to Staphylococcus Aureus Treated With DAIR.
Acronym: PhagoDAIRI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phaxiam Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-004469-11
Record Dates: First submitted 2022-04-27; First posted 2022-05-11 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Infection of Total Hip Joint Prosthesis; Infection of Total Knee Joint Prosthesis
Keywords: Joint Infection; Staphylococcus aureus; Phagotherapy
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Intervention Model Description: This is a pilot, randomized, non-comparative, double-blind study in patients with knee or hip prosthetic joint infection (PJI) due to Staphylococcus aureus, with the indication of DAIR and Suppressive Antibiotics Therapy (SAT). A stratification will be performed on the affected area of arthroplasty: knee or hip and on study site.
Who Masked: Participant, Investigator
Masking Description: All persons will be blinded, except the pharmacist will be unmasking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacteriophages arm (Experimental): 1 mL (PP1493 or PP1815) or 2 mL (PP1493 and PP1815) of suspension of bacteriophages diluted in solution of NaCl 0,9% at the end of DAIR procedure.
  Interventions: Biological: Anti-Staphylococcus aureus Bacteriophages
- Control Arm (Placebo Comparator): One local administration of NaCl 0,9% solution is administered at the end of the DAIR procedure.
  Interventions: Biological: Anti-Staphylococcus aureus Bacteriophages

INTERVENTIONS:
Biological: Anti-Staphylococcus aureus Bacteriophages — Single intra-articular injection

SUMMARY:
Pilot non comparative study assessing the clinical control of infection of DAIR + SAT +NaCl and DAIR + SAT + Phages anti-Staphylococcus aureus in patients with Staphylococcus aureus Prosthetic Joint Infection with an indication of DAIR + SAT.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years
2. Staphylococcus aureus monomicrobial knee or hip PJI ˃3 months after prosthesis implantation with clinical signs of infection and with indication of DAIR with direct closure and Suppressive Antibiotics Therapy (SAT)
3. Staphylococcus aureus only in joint fluid within 6 months before randomization or in case of relapse of infection under antibiotics therapy after a DAIR performed within 6 months before pre-inclusion visit
4. Without preoperative diagnosis of superinfection due to another pathogen
5. Phagogram displaying the susceptibility of the strain to at least one of the phages.
6. Patient with a life expectancy of 2 years and more as determined by the principal investigator
7. Females of childbearing potential/Sexually active males with partner of childbearing potential: commitment to consistently and correctly use an acceptable method of birth control (oral, transdermal, systemic or implant contraception birth control, intrauterine devices) for 1 month after the last study drug administration
8. Females of non-childbearing potential: either surgically sterilized or at least 1 year postmenopausal (amenorrhea duration at least 12 months)
9. Negative pregnancy test

Exclusion Criteria:

1. Early Staphylococcus aureus Prosthesis Joint infection (˂3months after the prosthesis implantation)
2. Other germ found in culture of joint fluid sample
3. Phagogram displaying no susceptibility of the strain to anti-Staphylococcus aureus bacteriophages
4. Patients with ASA score ≥ 4
5. Severe sepsis or Septic shock or hemodynamic instability
6. Patients with an indication to prosthesis replacement or amputation
7. Immunosuppressed patients
8. ALT or AST > 5 x ULN, creatinine > 1.53 mg/dl in men and > 1.24 mg/dl in women
9. Known allergic reactions to components of phages products
10. Medical history which in the opinion of the investigator would mean that the patient is unsuitable for participation in the study
11. Patients who are pregnant or breastfeeding. Patients should not be enrolled if they plan to become pregnant during the treatment period and 1 month after the last administration of study drug
12. Women/Men refusing to use an effective contraception during 1 month after the last administration of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-12-16 (Estimated); Study Completion 2025-06-16 (Estimated)

PRIMARY OUTCOMES:
Clinical control of infection at week 12 visit | week 12 visit
  No Fever, no recurrence, no worsening of pain, no periarticular inflammatory and clinical infectious signs, no new surgical request, no Staphylococcus aureus detected in joint fluid.

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events | From the time of signing the informed consent form up to study end visit (Months 24)
  Incidence, severity and type of adverse events and serious adverse events
Clinical laboratory tests | From the time of signing the informed consent form up to study end visit (Months 24)
  Number of participants with abnormal clinical laboratory tests
Physical examination | From the time of signing the informed consent form up to study end visit (Months 24)
  Number of participants with clinically abnormal physical examination findings
Clinical control of infection after Week 12 visit | Month 6, Month 12, Month 18 and Month 24.
  No Fever, no recurrence, no worsening of pain, no periarticular inflammatory and clinical infectious signs, no new surgical request, no Staphylococcus aureus detected in joint fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Pr Tristan Ferry, Lyon, France

IPD SHARING:
Plan to Share IPD: No